CLINICAL TRIAL: NCT06865248
Title: Investigation of Psychometric Properties of the Turkish Version of the Modified Mini Mental State Examination in Typically Developing Children and Children With Neurodevelopmental Disorders
Brief Title: Psychometric Properties of the Turkish Version of the Modified Mini Mental State Examination
Status: Not yet recruiting | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Other Study IDs: ETK000000001
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Children; Neurologic Disorder; Cerebral Palsy; Down Syndrome; Healthy
MeSH Terms: conditions — Nervous System Diseases; Cerebral Palsy; Down Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One of the most commonly used screening tests for the mental status of adults is the Standardized Mini Mental State Examination (MMSE). The MMSE is designed to screen for cognitive dysfunction, assess the severity of impairments, and identify changes over time. In the country of the researchers, the Turkish adaptation of the MMSE for children has not been done and the validity and reliability of the Turkish version has not been demonstrated. This paper aims to investigate the pschiatric features of the MMSE for Turkish pediatric population.

DETAILED DESCRIPTION:
Cerebral Palsy progresses with neurosensory, behavioral and cognitive disorders, especially restrictive adaptive behaviors, and a wider range of symptoms and functional disorders (1). Cognitive functions are all the brain functions required to receive stimuli from the outside and inside, select stimuli, create responses and coordinate with the environment (2). During childhood, cognitive functions can be negatively affected by many diseases, conditions or health problems. Evaluation of cognitive functions is important to determine whether cognitive abilities deviate from normal, to treat and monitor them. For this reason, many different tests are used in different age groups. These are; Montreal cognitive assessment (MoCA), Raven matrices, Wechsler adult intelligence scale (WAIS), Rey-identity and response memory test, Bender visual motor perception test, Delis-kaplan verbal reasoning test (D-KEFS), Stroop Test and Verbal memory tests are some of them. These tests are usually specific to their fields and may require trained professionals for long application periods. One of the most commonly used screening tests for adults is the Standardized Mini Mental State Examination (MMSE). The MMSE is designed to screen for cognitive dysfunctions, assess the severity of the disorders, and determine changes over time. The MMSE was developed by Folstein and colleagues (3) to rapidly assess cognitive functions. It consists of five sections: orientation, registration, attention and calculation, recall, and language, and is scored out of 30 points. Some of the existing screening tools used in childhood are limited in their use due to their reliance on parental reports, unknown correlations with general intelligence, the need for motor skills, literacy, and lack of sensitivity to developmental change. Therefore, it has been determined that there is a need for low-cost, rapidly administerable short cognitive screening tools that will allow rapid assessment of a wide range of cognitive domains in childhood. In this context, pediatric versions of the MMSE have begun to be used in various countries, such as Australia (4), India (5), Niger (6), Spain (7), and the USA (8). However, the psychometric properties of the MMSE in children with CP have only been reported in Brazil by Moura et al. (9). The Turkish adaptation of the MMSE has not been made for children and the validity and reliability of the Turkish version has not been demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5-18,
* Children diagnosed with neurodevelopmental disorders (Attention Deficit and Hyperactivity Disorder, Specific Learning Disorder, Autism Spectrum Disorder, Motor Disorders (Spastic SP)
* Children who can understand and apply Turkish commands

Exclusion Criteria:

Those with have serious hearing and speech problems

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged between the years of 5 and 18 who were diagnosed with neurodevelopmental disorders (Attention Deficit and Hyperactivity Disorder, Specific Learning Disorder, Autism Spectrum Disorder, Motor Disorders (Spastic SP)
Sampling Method: Probability Sample
Enrollment: 397 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Modified Mini Mental State Examination | at baseline and on the 7th day from the baseline
  Its scoring is between 0-12. For attention; it consists of 2 sub-items as counting forward and backward. The total score is between 0-7. For sensory perception; the child will be asked to name 3 known objects (pen, watch, glasses). Its scoring is between 0-3. For recall; the child will be asked to show and explain the previous 3 objects (pen, watch, glasses). Its scoring is between 0-3. For language; first, the child will be asked to name the 5 determined body parts (hand, foot, knee, nose, ear), second, they will be asked to carry out a 3-stage command, third, they will be asked to repeat a tongue twister, fourth, they will be asked to read and apply the shown text (close their eyes), fifth, they will be asked to write their name and finally they will be asked to draw the shown shape. Scoring ranges from 0 to 12. The highest score that can be obtained from the Modified MMSE is 37. Application time is between 8-15 minutes.

SECONDARY OUTCOMES:
Colored Progressive Matrices Test (RPM) | at baseline and on the 7th day from the baseline
  In each matrix consisting of meaningless shapes in parts called A, AB and B, there is a shape with a missing part. It will be asked to find the correct one from the 6 options that complete the missing part in the bottom part. It will receive 1 point for each correct answer.
Functional Independence Measure for Children (WeeFIM) | at baseline and on the 7th day from the baseline
  It consists of 6 sections including self-care (eating, washing hands and face, brushing teeth, toileting, bathing and dressing), sphincter control (bladder and bowel habits), transfer (transfer to toilet, shower and chair), locomotion (walking, crawling, going up and down stairs), communication (understanding and expressing) and social status (social relationships, problem solving and memory) and contains a total of 18 items. The family will be asked to score each item in these sections from 1 to 7 according to whether the individual received help while performing the function, whether he/she did it on time or whether an assistive device was required. The "Self-Care" subscale will be used in this study. The child's level of independence in daily life will be recorded by asking 6 questions here.

CONTACTS AND LOCATIONS:
Overall Officials: Emine HANDAN TÜZÜN, Prof., Study Director — Eastern Mediterranean University
Locations (1):
- Zehra Güçhan Topcu, Famagusta, Cyprus